# COMPARISON OF TWO TECHNIQUES FOR THE TREATMENT OF CARPAL TUNNEL SYNDROME. RANDOMIZED CLINICAL TRIAL

ID: NCT05468814

Date: January 27, 2022

#### STUDY PROTOCOL

## **Objectives**

To determine if the incidence of postoperative pillar pain is lower for either of the two surgical techniques being studied after 3 weeks and 6 months of follow-up Secondary, to check if the post-surgical grip strength, pinch strength and Borton Carpal Tunnel Questionnaire (BCTQ) score are better for either of the two surgical techniques

#### Design

Randomised clinical trial.

#### Methods

### Study variables

| Signs of compression of the median nerve: pain and paresthesias in the first three |
|---|
| fingers and radial edge of the fourth finger, nocturnal paresthesias, thenar muscle |
| atrophy, loss of opposition of the thumb. Durkan, Phalen, Tinel signs. |
| Pillar pain: pain/sensation of allodynia in the area of the thenar and/or hypothenar |
| eminence, hyperalgesia in the scar, pain when supporting the heel of the hand, |
| dysesthesia at rest. |
| Questionnaire: BCTQ (Boston Carpal Tunnel Syndrome Questionnaire). |
| Grip strength and pinch strength with specific dynamometers |

#### *Inclusion criteria*

- 1) Age > 18 years
- 2) Moderate-severe carpal tunnel syndrome
- 3) Symptoms that hinder the patient's daily activities
- 4) Have performed a correct conservative treatment without success

### Exclusion criteria

- 1) Previous carpal tunnel syndrome surgery
- 2) Traumatic or congenital sequelae of the hand
- 3) Unable to understand the process and the tests to be performed

#### Design

The follow-up process was carried out in three visits (3 weeks and 6 months after surgery).

In the **pre-surgery visit**, we carried out: patient screening and recruitment, patient information and obtaining informed consent process, application of the **inclusion and exclusion criteria**, medical history and physical examination of the hand to reach the **clinical and exploratory diagnosis of carpal tunnel syndrome**, obtaining baseline values from the **BCTQ questionnaire**, obtaining baseline **grip** and **pinch strength** values. After that, patients were **randomly assigned** to one of two treatment groups. Once included in each study group, the specific **surgical operation** was carried out. Finally, in the **post-surgery visits (3 weeks and 6 months** post-surgery), we evaluated: clinical and

examination of the median nerve compression clinic, presence or not of **pillar pain**, post-operative BCTQ values and grip and pinch strengths.

### STATISTICAL ANALYSIS PLAN (SAP)

To carry out the sample homogeneity study, the statistical Student t-tests for the quantitative variables and chi-square for the qualitative variables were used. For the analysis of the qualitative variables the chi-square statistical test was used. Mixed ANOVA was used using the patient as a random effect and using the visit and surgical technique as a fixed effect to analyse the absolute change in grip and pinch strength and the BCTQ score after 3 weeks and 6 months after surgery.

As for the data analysis, two new variables were created for the quantitative variables: the <u>absolute change</u> in grip strength, in pinch strength and in the BCTQ score and the <u>relative change</u> therein, performed by an absolute and percentage calculation (respectively) of the difference between values after 3 weeks from baseline and values after 6 months from baseline; i.e., comparing each patient with themself calculating the variation in these variables throughout the follow-up.

Finally, the Student's t-test was used to study the absolute and relative change in the grip and pinch strength and BCTQ values.